CLINICAL TRIAL: NCT00002391
Title: A Double-Blind, Randomized, Multicenter Trial to Evaluate the Safety and Efficacy of the Combination of 1592U89/Zidovudine (ZDV)/Lamivudine (3TC) Versus the Combination of Zidovudine (ZDV)/Lamivudine (3TC) in HIV-1 Therapy-Experienced Pediatric Patients.
Brief Title: The Safety and Effectiveness of Zidovudine Plus Lamivudine, Used With and Without 1592U89, in HIV-1 Infected Children Who Have Taken Anti-HIV-1 Drugs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 238L; CNAA3006
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-11

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Therapy, Combination; Zidovudine; Lamivudine; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load; Child Development; abacavir
MeSH Terms: conditions — HIV Infections | interventions — abacavir; Lamivudine; Zidovudine

INTERVENTIONS:
Drug: Abacavir sulfate
Drug: Lamivudine
Drug: Zidovudine

SUMMARY:
To compare the safety, tolerance, durability of the viral load response and the antiviral activity of the 1592U89/zidovudine(ZDV)/lamivudine (3TC) regimen vs. ZDV/3TC regimen. To determine the clinical efficacy of the two regimens as measured survival, disease progression, weight growth velocity, and neuropsychological or neurological changes. To assess the development of viral resistance and relative pharmacokinetics associated with each regimen.

DETAILED DESCRIPTION:
Patients are randomized to receive blinded treatment with ZDV/3TC alone or in combination with 1592U89, orally for 16 weeks. If after the 16-week period certain criteria are met, patients may have the option to switch to open-label treatment for the remainder of the study period.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Intravenous immunoglobulin G, erythropoietin, G-CSF and GM-CSF.
* Opportunistic infection prophylaxis.

Patients must have:

* HIV-1 infection documented by:

< 18 months of age:

* one positive viral test culture and one other positive viral test (culture, PCR, p24 antigen, or Immune Complex Dissociation p24 antigen) on two different specimens.

>= 18 months of age:

* two positive viral tests as stated above, one or both of which may be determined by a federally documented ELISA and confirmed by Western blot or Indirect Fluorescent Antibody test.
* Any of the CDC Categories:
* 1, 2, 3, and N, A, B, and C of the 1994 Revised Classification System for HIV Infection in Children Less than 13 Years of Age.
* CD4+ count >= 15% within 14 days prior to study drug administration.
* No active or ongoing AIDS-defining opportunistic infection that precludes absorption of study drug or observation of a study parameter.
* Signed, informed consent from parent or legal guardian for patients under 18 years of age.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Serious bacterial infection that precludes absorption of study drug or observation of a study parameter.
* Documented hypersensitivity to a nucleoside analog.
* Co-enrollment in certain opportunistic infection protocols is not exclusionary if approval is obtained.
* Malignancy.
* Life-threatening infection or other chronic disease that may compromise patient safety.
* Grade 3/4 clinical or laboratory toxicity or current grade 2 or higher pancreatic amylase or lipase toxicity as defined by the ACTG Toxicity Tables within 14 days prior to study entry.

Concurrent Medication:

Excluded:

* Other anti-HIV therapy.
* Probenecid.
* Biologic response modifier (unless listed under included concurrent medication) and megestrol acetate.
* Human growth hormone.
* Immunomodulators and cytotoxic chemotherapeutic agents.
* Systemic corticosteroids > 14 days without approval.
* Investigational agents.

Concurrent Treatment:

Excluded:

Radiation therapy.

Patients with the following prior conditions are excluded:

* History of clinically relevant pancreatitis or hepatitis within the past 6 months.
* Participation in a vaccine trial.

Prior Medication:

Excluded:

* Protease inhibitor therapy within 2 weeks prior to randomization.
* Interleukins or interferons within 30 days prior to study drug administration.
* Investigational drugs within 14 days prior to randomization.
* HIV vaccine dose within past 30 days.

Required:

> 12 weeks prior antiretroviral therapy and unchanged therapy 12 weeks prior to screening.

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child

CONTACTS AND LOCATIONS:
Locations (30):
- United States (30):
  - Univ Alabama - Birmingham / Dept of Pediatrics / UAB Station, Birmingham, Alabama
  - Children's Hosp Los Angeles, Los Angeles, California
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - Children's Diagnostic Treatment Ctr, Fort Lauderdale, Florida
  - Univ of Florida - Gainesville / Infectious Dis & Immun, Gainesville, Florida
  - Univ of Miami / Fox Cancer Research Ctr, Miami, Florida
  - Arnold Palmer Hosp for Women and Children, Orlando, Florida
  - Pediatric Special Immunology Clinic / HRS / PBC PHU, Riviera Beach, Florida
  - Univ of South Florida All Children's Hosp, St. Petersburg, Florida
  - Dr Patricia Emmanuel, Tampa, Florida
  - Mt Sinai Hosp Med Ctr / Dept of Pediatrics, Chicago, Illinois
  - Tulane Univ Med School, New Orleans, Louisiana
  - Univ of Minnesota Med School, Minneapolis, Minnesota
  - UMDNJ / Division of Allergy Immunology & Infectious Diseases, Newark, New Jersey
  - PACT Program, Buffalo, New York
  - North Shore Univ Hosp / Pediatric Immunology, Great Neck, New York
  - Schneider Children's Hosp, New Hyde Park, New York
  - New York Hosp - Cornell / Program for Children with AIDS, New York, New York
  - St Luke's - Roosevelt Hosp Ctr, New York, New York
  - SUNY Health Ctr at Stony Brook / Pediatric Infectious Dis, Stony Brook, New York
  - SUNY Health Sciences Ctr at Syracuse / Dept of Pediatrics, Syracuse, New York
  - Bronx Lebanon Hosp Ctr / Dept of Pediatrics, The Bronx, New York
  - Univ of North Carolina / Pediatric Infectious Diseases, Chapel Hill, North Carolina
  - Duke Univ Med Ctr / Pediatrics Dept / Infec Dis, Durham, North Carolina
  - The Children's Med Ctr / Division of Infectious Dis, Dayton, Ohio
  - Med Univ of South Carolina, Charleston, South Carolina
  - Children's Med Ctr of Dallas / ARMS Clinic, Dallas, Texas
  - Cook's Ft Worth Children Med Ctr / Pediatric Inf Dis, Fort Worth, Texas
  - Univ of Texas Health Sciences Ctr, San Antonio, Texas
  - Eastern VA Med Sch / Children's Hosp of the King's Daughters, Norfolk, Virginia